CLINICAL TRIAL: NCT06577961
Title: Study on the Efficacy and Safety of Vorolanib Combined With Cadonilimab in the Treatment of Untreated Advanced RCC Patients
Brief Title: Vorolanib Combined With Cadonilimab in the Treatment of Untreated Advanced RCC Patients
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Xiongjun Ye, Chief Physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-FL-IV008
Record Dates: First submitted 2024-07-11; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Kidney Cancer; RCC; Renal Cell Carcinoma
Keywords: Kidney Cancer; RCC; Renal Cell Carcinoma; vorolanib Combined with Cadonilimab
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — vorolanib

STUDY DESIGN:
Intervention Model Description: Vorolanib combined with cadonilimab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Vorolanib combined with cadonilimab
  Interventions: Drug: Vorolanib; Drug: cadonilimab

INTERVENTIONS:
Drug: Vorolanib — stage Ⅰ：Vorolanib 200mg QD stage Ⅱ：Vorolanib RP2D QD
  Other Names: CM082
Drug: cadonilimab — stageⅠ：cadonilimab 10mg/kg Q3W stageⅡ：cadonilimab 10mg/kg Q3W
  Other Names: AK104

SUMMARY:
Evaluate the efficacy and safety of vorolanib combined with cadonilimab in the treatment of untreated advanced RCC patients.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, phase I/II single-arm trial, aiming to enroll 37 untreated patients with advanced or metastatic ccRCC to receive vorolanib combined with cadonilimab treatment, and to perform CTC/ctDNA testing on subjects.

In the phase I dose exploration phase, a 3+3 dose escalation method is used to explore the safety of vorolanib at the standard dose combined with cadonilimab within one treatment cycle, and to determine the dose.

In the phase II trial phase, the dosage of vorolanib is determined by the optimal tolerated dose found in the phase I trial, while cadonilimab is combined for treatment.

Patients need to be evaluated for efficacy and safety after every 2 treatment cycles (within ±3 days at the end of each cycle), and continue treatment until disease progression, intolerable toxicity, or completion of the prescribed treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in this study, willing and able to comply with and sign the informed consent form;
2. Histologically confirmed clear cell renal cell carcinoma;
3. Advanced (not suitable for curative surgery or radiation therapy) or metastatic (AJCC Stage IV) RCC;
4. No prior systemic treatment for RCC, except for the following situations:

   a) For completely resectable renal cell carcinoma, having received one type of adjuvant or neoadjuvant treatment, if the treatment does not include drugs targeting VEGF or VEGFR, and recurrence occurs at least 6 months after the last adjuvant or neoadjuvant treatment;
5. Confirmed to have at least one measurable lesion according to RECIST 1.1 criteria;
6. KPS score ≥ 70;
7. Expected survival time of more than 3 months;
8. Aged 18-75 years;
9. Good function of major organs and sufficient hematology, meeting the following criteria:

   Absolute neutrophil count (ANC) ≥ 1500 cells/μL (no granulocyte colony-stimulating factor support within 2 weeks before Cycle 1, Day 1) Platelet count (PLT) ≥ 80 × 10^9/L. WBC count ≥ 2500/μL without G-CSF, ≤ 15000/μL Lymphocyte count ≥ 500/μL Hemoglobin ≥ 9.0 g/dL (Cycle 1), not dependent on erythropoietin, and no transfusion of concentrated red blood cells (pRBC) in the past 2 weeks Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP) ≤ 3 times the upper limit of normal (ULN) (liver metastasis ≤ 5 times ULN). If the patient has bone metastasis, ALP ≤ 5 times ULN.

   Serum bilirubin ≤ 1.5 × ULN. Patients with known Gilbert's syndrome can be enrolled if serum bilirubin level ≤ 3 times ULN.

   Serum albumin ≥ 2.8 g/dL Creatinine ≤ 2.0 × ULN or calculated creatinine clearance rate ≥ 30 mL/min. Urine protein/creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.2 mg/mmol)
10. For women who are not menopausal (amenorrhea for 12 months) or surgically sterile (without ovaries and/or uterus): agree to use two appropriate methods of contraception, including at least one method with an annual failure rate of ≥ 1%.
11. Sexually active subjects of childbearing potential and their partners must agree to use medically recognized contraceptive methods during the study and for 5 months after the last dose of study treatment for women and 7 months for men (e.g., barrier methods, including male condoms, female condoms, or diaphragms coated with spermicidal gel).
12. Female subjects of childbearing potential must not be pregnant at screening. Women of childbearing potential are defined as premenopausal women who can become pregnant (i.e., women who have had any menstrual signs in the past 12 months, except for those who are surgically sterile as mentioned above).However, women who have been amenorrheic for 12 months or longer are still considered to have childbearing potential if the amenorrhea is likely due to previous chemotherapy, anti-estrogens, low body weight, ovarian suppression, or other reasons.

Exclusion Criteria:

1. Received any systemic treatment for RCC, unless the investigator can provide evidence that the subject has been randomly assigned to the placebo group;
2. Central nervous system metastasis;
3. Active malignant tumor in the past 24 months (except for renal cell carcinoma, skin basal cell carcinoma or squamous cell carcinoma that has been clearly treated, as well as cervical or bladder carcinoma in situ). Participants with a history of localized and low-risk prostate cancer who have received curative treatment and have not had a prostate-specific antigen (PSA) recurrence in the past 5 years may participate in the study;
4. Received prior radiotherapy within 21 days before the start of study treatment (palliative radiotherapy for bone lesions is allowed, provided it is completed at least 2 weeks before the start of study treatment);
5. Currently participating in another study or received study drugs within 4 weeks before the start of study treatment.
6. Receiving live vaccines within 30 days after the planned start of study treatment (first cycle/day 1). Live vaccines include but are not limited to measles, mumps, rubella, varicella/zoster (chickenpox), yellow fever, rabies, BCG, and typhoid vaccines. Injectable seasonal influenza vaccines are generally inactivated virus vaccines and are allowed; however, intranasal influenza vaccines are attenuated live vaccines and are not allowed.
7. Participants with proteinuria > 1+ on urine dipstick test will undergo a 24-hour urine collection for quantitative assessment of proteinuria. Participants with urinary protein ≥ 1g/24h will not be eligible.
8. Fasting total cholesterol > 300 mg/dL (or 7.75 mmol/L) and/or fasting triglyceride level 2.5 times the upper limit of normal (ULN). Note: These participants can be included after lipid-lowering treatment.
9. Uncontrolled diabetes defined as fasting blood glucose > 1.5 times the upper limit of normal. Note: These participants can be included after hypoglycemic treatment.
10. Uncontrolled hypercalcemia (≥ 1.5 mmol/L ionized calcium or Ca ≥ 12 mg/dL or corrected serum calcium ≥ ULN) or symptomatic hypercalcemia requiring continued bisphosphonate treatment or denosumab.
11. QTc interval prolongation to > 480 ms.
12. Participants who have not fully recovered from any toxicity and/or complications caused by major surgery before starting treatment.
13. Malabsorption, gastrointestinal anastomosis, or any other condition that may affect the absorption of study drugs.
14. Clinically significant hematuria, vomiting blood, or coughing up blood > 0.5 teaspoon (2.5 ml) within 12 weeks before the first dose, or other significant bleeding history (such as pulmonary hemorrhage).
15. Significant cardiovascular impairment within 12 months after the first dose of study drug: history of congestive heart failure New York Heart Association class II or higher, unstable angina, myocardial infarction, cerebrovascular accident, or arrhythmia related to hemodynamic instability. The following conditions are also excluded: left ventricular ejection fraction (LVEF) below the institutional normal range determined by gated blood pool scan or echocardiogram.
16. Active infection (any infection requiring systemic treatment).
17. Positive for human immunodeficiency virus (HIV).
18. Active hepatitis B or C.
19. Known history of interstitial lung disease or any evidence.
20. History of (non-infectious) pneumonia requiring steroids, or currently suffering from pneumonia.
21. Diagnosed with immunodeficiency or receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days before the first study treatment. Physiological doses of corticosteroids (up to 10 mg/day prednisone or equivalent) can be used during the study period.
22. Active autoimmune disease requiring systemic treatment within the past 2 years (excluding psoriasis). Alternative therapies (such as thyroid hormones, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency) are not considered forms of systemic treatment.
23. Breastfeeding or pregnant women at screening or baseline.
24. Fertile women who do not agree to use highly effective contraceptive methods throughout the study period and for 120 days after the end of the study.
25. Men who have not successfully undergone vasectomy (diagnosed with azoospermia) and do not agree to use condoms/spermicides from the first dose of study treatment until 120 days after the last dose of study treatment, unless they practice abstinence.
26. Known intolerance to any study drug (or any excipient).
27. Participants who have received allogeneic tissue/solid organ transplantation.
28. Patients requiring pain medication must be on a stable treatment regimen at the start of the study.
29. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage (monthly or more frequently).
30. Uncontrolled hypertension defined as persistent blood pressure (BP) > 150 mmHg systolic or > 100 mmHg diastolic.
31. Unable to swallow tablets or capsules.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-08-31 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate assessed by RECIST 1.1 | 12 months
  ORR, per RECIST 1.1 calculated as the proportion of patients with a best overall response defined as complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Progression Free Survival assessed by the investigator | 24 months
  PFS, defined as time from study drug administration to progression or death due to any cause.disease progression (PD) or death due to any reason. Imaging assessment is based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | 24 months
  During the AE reporting period specified in the protocol, collect all AEs (including SAEs) and record them in the CRF form.
Overall Survival | 24 months
  OS, defined as the time from study drug administration until the date of death due to any cause.
Disease Control Rate | 12 months
  DCR, defined as proportion of complete response, partial response, and disease stabilization to the proportion of patients with evalueable tumors.
12 months Progression Free Survival Rate | 12 months
  The progression-free survival rate is evaluated for all enrolled patients from the start of the first treatment to 12 months.
12 months Overall Survival Rate | 12 months
  Assess the overall survival rate for all enrolled patients from the start of the first treatment to 12 months.
24 months Overall Survival Rate | 24 months
  Assess the overall survival rate for all enrolled patients from the start of the first treatment to 24 months.
Health-related quality of life | 24 months
  Use the EORTC Quality of Life Questionnaire Core 30 (QLQ-C30) to conduct a questionnaire survey on subjects.

OTHER OUTCOMES:
Circulating Tumor Cell / circulating tumor DNA | It is anticipated that blood tests will be conducted on patients before medication, 42±3 days after medication, and within 7 days following disease progression.
  Exploration of biomarkers with potential clinical value for the clearance of circulating tumor cells/DNA

CONTACTS AND LOCATIONS:
Overall Officials: xiongjun YE, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences

IPD SHARING:
Plan to Share IPD: No